CLINICAL TRIAL: NCT01924338
Title: Validierung Der Bestimmung Der Gewebedicke Mit Hilfe Von Licht im Infrarotbereich
Brief Title: Validation of a Method to Measure Soft Tissue Thickness Using Near Infrared Laser Light
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Floris Ernst (Other)
Collaborators: Varian Medical Systems (Industry); University of Luebeck (Other)
Responsible Party: Sponsor-Investigator, Dr. Floris Ernst, Senior Research Associate, University of Luebeck
Organization: University of Luebeck (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROB-NIRMR-001
Record Dates: First submitted 2013-08-12; First posted 2013-08-16 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Cranial Soft Tissue
Keywords: Patient; localisation; in cranial; radiation; therapy; thickness of
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Skin types I and II (Experimental): Volunteers classified as skin types I and II according to the Fitzpatrick Scale
  Procedures: dental cast creation, MRI scan, laser scan
  Interventions: Device: MRI scan; Device: Laser scan; Procedure: Dental cast creation
- Skin type III (Experimental): Volunteers classified as skin type III according to the Fitzpatrick Scale
  Procedures: dental cast creation, MRI scan, laser scan
  Interventions: Device: MRI scan; Device: Laser scan; Procedure: Dental cast creation
- Skin type IV (Experimental): Volunteers classified as skin type IV according to the Fitzpatrick Scale
  Procedures: dental cast creation, MRI scan, laser scan
  Interventions: Device: MRI scan; Device: Laser scan; Procedure: Dental cast creation
- Skin types V and VI (Experimental): Volunteers classified as skin types V and VI according to the Fitzpatrick Scale
  Procedures: dental cast creation, MRI scan, laser scan
  Interventions: Device: MRI scan; Device: Laser scan; Procedure: Dental cast creation

INTERVENTIONS:
Device: MRI scan — Acquisition of a high-resolution MRI scan (0.15 x 0.15 x 1.0 mm³) aligned with the AC-PC (anterior commissure-posterior commissure) line
Device: Laser scan — A near-infrared laser scan of the subject's forehead is acquired
Procedure: Dental cast creation — A dental cast made of PMMA (polymethyl methacrylate) of the subject's maxilla is created

SUMMARY:
The study is intended to verify a newly developed method to measure the thickness of cranial soft tissue. In the study, a high-resolution MRI scan is used as ground truth for a laser scan of the forehead. The laser scan is acquired point by point with a prototype scanning unit developed at the University of Luebeck's Institute for Robotics.

The measured tissue thickness using the near-infrared scanning approach is validated against the ground truth obtained by the MRI scan. The average accuracy of the reconstruction method is then computed over all subjects from the individual study arms.

The required laser intensity and exposure time as well as the achieved measurement accuracy is evaluated with respect to the different skin types of the test subjects. Correlation between these features and the skin type according to the Fitzpatrick scale will be computed.

For 1/3 of the subjects, the laser and MRI scans are repeated after 2 and 8 weeks. The results of the scans are compared and time dependency is analysed.

ELIGIBILITY:
Inclusion Criteria:

* male and female adults
* variations in skin type (at least 10 subjects with skin types I & II, at least 2 subjects with skin type III, at least 3 subjects with skin type IV, at least 3 subjects with skin types V & VI)
* optional: availability of high-resolution CT or CBCT (cone-beam CT) scan of the forehead

Exclusion Criteria:

* allergies or intolerances against ABS (acrylonitrile butadiene styrene), PMMA (polymethyl methacrylate) or alginate
* elevated light sensitivity of the skin
* exclusion criteria for MRI (claustrophobia, motoric disorders, tattoos, body piercings, metallic implants in the skull, epilepsy, cardiac pacemakers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Average accuracy of tissue thickness measurement method [mm] | up to 6 months

SECONDARY OUTCOMES:
System dependency on skin color - required intensity | up to 6 months
  Correlation between skin types (according to the Fitzpatrick scale) and the outcome (required laser intensity [mW])
Long-term stability of measured features - accuracy | up to 8 months
  Change in measurement accuracy [mm]
Long-term stability of measured features - required intensity | up to 8 months
  Change in required laser intensity [mW]
Long-term stability of measured features - required exposure time | up to 8 months
  Change in required exposure time [ms]
System dependency on skin color - accuracy | up to 6 months
  Correlation between skin types (according to the Fitzpatrick scale) and the outcome (accuracy of tissue thickness measurement [mm])
System dependency on skin color - exposure time | up to 6 months
  Correlation between skin types (according to the Fitzpatrick scale) and the outcome (required exposure time [ms])

CONTACTS AND LOCATIONS:
Overall Officials: Floris Ernst, PhD, Principal Investigator — University of Luebeck
Locations (2):
- Germany (2):
  - Clinic for Maxillofacial Surgery of the University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - University of Luebeck, Institute for Robotics, Lübeck, Schleswig-Holstein

REFERENCES:
- [Background] Wissel T, Bruder R, Schweikard A, Ernst F. Estimating soft tissue thickness from light-tissue interactions--a simulation study. Biomed Opt Express. 2013 Jun 14;4(7):1176-87. doi: 10.1364/BOE.4.001176. Print 2013 Jul 1. PMID 23847741